CLINICAL TRIAL: NCT02025764
Title: The Clinical Feature of the Exposed Vessels in Ulcer Base Over Time After Prophylactic Argon Plasma Coagulation in Colonic Endoscopic Mucosal Resection
Brief Title: The Clinical Feature of Ulcer Base Over Time After Prophylactic Argon Plasma Coagulation in Colonic EMR
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Yunho Jung, Assistant Professor, Soonchunhyang University Hospital
Other Study IDs: SCHCA_IRB_2013-56
Record Dates: First submitted 2013-12-10; First posted 2014-01-01 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Gastrointestinal Hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

SUMMARY:
The prophylactic APC right after colonic EMR doesn't mean the complete coagulation of visible vessel because of injection material.

The aim of this study was to evaluate the clinical feature of the visible vessels in ulcer base over time after prophylactic APC in colonic EMR.

DETAILED DESCRIPTION:
The prophylactic Argon plasma coagulation (APC) of non-bleeding visible vessels seems not to have an additional advantage in the prevention of delayed post polypectomy bleeding in recently studies. However, immediate APC after endoscopic mucosal resection (EMR) may not mean the complete coagulation of exposed vessels because of injection material. The aim of this study was to evaluate the clinical feature of the exposed vessels in ulcer base over time after prophylactic APC in colonic EMR. Methods: This study was designed as a prospective study. Investigators excluded diminutive polyp, large polyp (> 2cm), long stalk pedunculated polyp, and clear ulcer base after EMR. Between August 2013 and May 2014, patients who were enrolled underwent prophylactic APC for non-bleeding visible vessels after colonic endoscopic mucosal resection. After checking the complete coagulation of visible vessels, the numbers of visible vessel group were counted by lap of time such as 1, 3, 5, and 7 min in ulcer base.

ELIGIBILITY:
Inclusion Criteria:

* Underwent prophylactic APC for non-bleeding visible vessels after colonic endoscopic mucosal resection.

Exclusion Criteria:

* Diminutive polyp, large polyp (> 2cm), long stalk pedunculated polyp, and clear ulcer base after EMR.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Between August 2013 and May 2014, patients who were enrolled underwent prophylactic APC for non-bleeding visible vessels after colonic endoscopic mucosal resection.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
underwent prophylactic APC for non-bleeding visible vessels after colonic endoscopic mucosal resection. After checking the complete coagulation of visible vessels, the numbers of visible vessel group were counted in ulcer base. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Yunho Jung, Master, Principal Investigator — Soo Chun Hyang University Hospital Cheonan
Locations (1):
- Soon Chun Hyang University Hospital Cheonan, Cheonan, Chungcheonam-do, South Korea